CLINICAL TRIAL: NCT03387982
Title: Post Procedural Pain Assessment in Patients Undergoing Balloon Cryotherapy Compared to Radiofrequency Ablation (RFA) for Dysplastic Barrett's: A Prospective Study
Brief Title: Balloon Cryotherapy vs. Radiofrequency Ablation Pain Study
Status: Completed | Type: Observational
Sponsor: Geisinger Clinic (Other)
Collaborators: Medical University of South Carolina (Other); Long Island Jewish Medical Center (Other); Pentax Medical (Industry); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Hashit Khara, Clinical Assistant Professor of Medicine; Director of Endoscopic and Translational Research, Geisinger Clinic
Other Study IDs: 2017-0363
Record Dates: First submitted 2017-11-23; First posted 2018-01-02 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Balloon Cryotherapy Treatment Group: Subjects will undergo endoscopic balloon cryotherapy for dysplastic Barrett's Esophagus as per standard of care. The treatment type (balloon cryotherapy vs RFA) is determined by the endoscopy physician at the time of the procedure and is based on several clinical factors including co-existing medical conditions, the anatomy of the esophagus, and the length and amount of tissue affected with Barrett's.
- RFA Treatment Group: Subjects will undergo radio frequency ablation treatment for dysplastic Barrett's Esophagus as per standard of care. The treatment type (balloon cryotherapy vs RFA) is determined by the endoscopy physician at the time of the procedure and is based on several clinical factors including co-existing medical conditions, the anatomy of the esophagus, and the length and amount of tissue affected with Barrett's.

SUMMARY:
Barrett's esophagus is a condition in which the normal lining of the lower esophagus is replaced with cells that predispose an individual to development of esophageal cancer. Treatment of Barrett's esophagus reduces the risk of progression to cancer. Treatment is provided endoscopically, via a variety of approved techniques including endoscopic mucosal resection, argon plasma coagulation, radiofrequency ablation (RFA), spray cryotherapy ablation and balloon cryotherapy ablation. A common side effect of ablation treatment is pain, thus making pain an important factor when discussing treatment options. It is speculated that balloon cryotherapy causes less pain than RFA but no head-to-head comparison trials exist to date. This multi-center, prospective cohort study aims to compare pre- and post-procedural pain for balloon cryotherapy versus RFA. Providing both patients and clinicians with data from a well-designed prospective study may help guide future physician/patient treatment discussions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dysplastic Barrett's esophagus (LGD and HGD) naïve to ablation therapy presenting for ablation
2. Age ≥ 18
3. Ability to sign informed consent

Exclusion Criteria:

1. Prior ablation treatment for Barrett's esophagus
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for treatment of Barrett's Esophagus.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Difference in pain quality immediately pre-procedure (Baseline) for subjects receiving Balloon Cryotherapy or Radiofrequency Ablation via the Pain Quality Assessment Scale (PQAS) | immediately before procedure
  Differences in PQAS scores between groups will be determined by using the t test or Wilcoxon test for continuous variables and the Fisher exact test for categorical variables. The Pain Quality Assessment Scale (PQAS) assesses distinct pain qualities associated with all types and categories of pain problems. The PQAS is a 20-item measure used to assess pain qualities associated with non-neuropathic pain. The PQAS asks respondents to rate the severity of each of 20 pain (quality and spatial) descriptor domains by using 0 to 10 numeric rating scales, in which 0 = "no pain" or "not [ descriptor/item]" and 10 = "the most [descriptor] pain sensation imaginable."
Difference in pain quality immediately post-procedure for subjects receiving Balloon Cryotherapy or Radiofrequency Ablation via the Pain Quality Assessment Scale (PQAS) | immediately post procedure
  Differences in PQAS scores between groups will be determined by using the t test or Wilcoxon test for continuous variables and the Fisher exact test for categorical variables. The Pain Quality Assessment Scale (PQAS) assesses distinct pain qualities associated with all types and categories of pain problems. The PQAS is a 20-item measure used to assess pain qualities associated with non-neuropathic pain. The PQAS asks respondents to rate the severity of each of 20 pain (quality and spatial) descriptor domains by using 0 to 10 numeric rating scales, in which 0 = "no pain" or "not [ descriptor/item]" and 10 = "the most [descriptor] pain sensation imaginable."
Difference in pain quality 2 days post-procedure for subjects receiving Balloon Cryotherapy or Radiofrequency Ablation via the Pain Quality Assessment Scale (PQAS) | 2 days post procedure
  Differences in PQAS scores between groups will be determined by using the t test or Wilcoxon test for continuous variables and the Fisher exact test for categorical variables. The Pain Quality Assessment Scale (PQAS) assesses distinct pain qualities associated with all types and categories of pain problems. The PQAS is a 20-item measure used to assess pain qualities associated with non-neuropathic pain. The PQAS asks respondents to rate the severity of each of 20 pain (quality and spatial) descriptor domains by using 0 to 10 numeric rating scales, in which 0 = "no pain" or "not [ descriptor/item]" and 10 = "the most [descriptor] pain sensation imaginable."
Difference in pain quality 1 week post-procedure for subjects receiving Balloon Cryotherapy or Radiofrequency Ablation via the Pain Quality Assessment Scale (PQAS) | 1 week post procedure
  Differences in PQAS scores between groups will be determined by using the t test or Wilcoxon test for continuous variables and the Fisher exact test for categorical variables. The Pain Quality Assessment Scale (PQAS) assesses distinct pain qualities associated with all types and categories of pain problems. The PQAS is a 20-item measure used to assess pain qualities associated with non-neuropathic pain. The PQAS asks respondents to rate the severity of each of 20 pain (quality and spatial) descriptor domains by using 0 to 10 numeric rating scales, in which 0 = "no pain" or "not [ descriptor/item]" and 10 = "the most [descriptor] pain sensation imaginable."
Difference in pain quality 4 weeks post-procedure for subjects receiving Balloon Cryotherapy or Radiofrequency Ablation via the Pain Quality Assessment Scale (PQAS) | 4 weeks post procedure
  Differences in PQAS scores between groups will be determined by using the t test or Wilcoxon test for continuous variables and the Fisher exact test for categorical variables. The Pain Quality Assessment Scale (PQAS) assesses distinct pain qualities associated with all types and categories of pain problems. The PQAS is a 20-item measure used to assess pain qualities associated with non-neuropathic pain. The PQAS asks respondents to rate the severity of each of 20 pain (quality and spatial) descriptor domains by using 0 to 10 numeric rating scales, in which 0 = "no pain" or "not [ descriptor/item]" and 10 = "the most [descriptor] pain sensation imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Harshit Khara, MD, Principal Investigator — Geisinger Clinic
Locations (4):
- United States (4):
  - Long Island Jewish Medical Center, Queens, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No